CLINICAL TRIAL: NCT06334705
Title: EGEA4: the 30-year Follow-up of the EGEA Study : Study of Markers of Cardiovascular Risk in Asthmatic and Non-asthmatic
Brief Title: EGEA4 THE 30 YEAR FOLLOW UP OF THE EGEA STUDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: APHP (Other); Hospices Civils de Lyon (Other); APHM (Unknown); University Hospital, Grenoble (Other); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C22-11; 2022-A02312- 41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-03-18; First posted 2024-03-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer EGEA4 Cohort
Keywords: Respiratory and cardiac health; Cohort; Epidemiology
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- participants can take part in any examinations they wish (Other)
  Interventions: Other: blood test, food collection, hair collection, calcium scan, etc.

INTERVENTIONS:
Other: blood test, food collection, hair collection, calcium scan, etc. — everything is specified during the phone call and in the consent form to be signed

SUMMARY:
Cardiovascular (CV) diseases affect 523 million people worldwide, and are the leading cause of death, accounting for over 18 million deaths (around 30% of all deaths) every year. CV diseases account for around 45% of all deaths in Europe, or around 140,000 deaths a year in France. Asthma is one of the main non-communicable diseases, with a significant societal and individual burden, particularly in subjects suffering from severe asthma. The prevalence of asthma worldwide has risen rapidly over the past five decades, and now affects 272 million people worldwide, representing a prevalence of around 3.6%.

Asthma is often associated with multimorbidity. Allergic rhinitis, chronic sinusitis, sleep apnea syndrome, gastro-oesophageal reflux disease, obesity and hormonal disorders are among the most common conditions associated with asthma. More recently, other chronic conditions linked to asthma have been suggested, including CV diseases.

Although data from the literature in recent years suggest that asthma is associated with an increased risk of major CV events, the underlying mechanisms remain poorly understood. In particular, it is not known whether asthma and CV disease share common etiological processes, such as anthropometric parameters, lifestyle, social, environmental and/or genetic factors, or whether CV disease is a direct consequence of certain features of asthma, such as systemic inflammation or asthma treatments.

Our study is based on the hypothesis that the risk of CV events is increased in patients with asthma, which is supported by a growing body of scientific data.However, it remains to be determined to what extent this increased risk is a consequence of asthma or is linked to shared risk factors between asthma and CV health.

We hypothesize that asthma, and more specifically adult and moderate-to-severe asthma, are associated with early markers of CV risk. Furthermore, by providing a better understanding of the mechanisms involved in this association, we hypothesize that EGEA_30years may help to disentangle and prioritize actionable levers of life-threatening cardiovascular comorbidities in asthma.

DETAILED DESCRIPTION:
Cardiovascular (CV) diseases, which include coronary heart disease and stroke, affect 523 million people worldwide and are the leading cause of death, accounting for over 18 million deaths (around 30% of all deaths) every year. CV diseases account for around 45% of all deaths in Europe, or around 140,000 deaths a year in France. Asthma is one of the main non-communicable diseases, with a significant societal and individual burden, particularly in subjects suffering from severe asthma. The worldwide prevalence of asthma has risen rapidly over the past five decades, and now affects 272 million people worldwide, representing a prevalence of around 3.6%, with considerable geographical variability.

Multimorbidity is common in asthma. Allergic rhinitis, chronic sinusitis, sleep apnea syndrome, gastroesophageal reflux disease, obesity and hormonal disorders are among the most common conditions linked to asthma.More recently, other chronic conditions linked to asthma have been suggested, including CV diseases.Although data from the literature in recent years suggest that asthma is associated with an increased risk of major CV events, the underlying mechanisms remain poorly understood. In particular, it is not known whether asthma and CV disease share common etiological processes, such as anthropometric parameters, lifestyle, social, environmental and/or genetic factors, or whether CV disease is a direct consequence of certain features of asthma, such as systemic inflammation or asthma treatments.

Our study is based on the hypothesis that the risk of CV events is increased in patients with asthma, which is supported by a growing body of scientific data.

However, it remains to be determined to what extent this increased risk is a consequence of asthma, or is linked to shared risk factors between asthma and CV health.We hypothesize that asthma, and more specifically adult and moderate-to-severe asthma, are associated with early markers of CV risk. Furthermore, by providing a better understanding of the mechanisms involved in this association, we hypothesize that EGEA_30years may help to disentangle and prioritize actionable levers of life-threatening cardiovascular comorbidities in asthma.

The main objectives of the EGEA4 study are:

1. to characterize the longitudinal association between asthma and cardiovascular (CV) risk assessed by the Framingham score,
2. study the association between asthma and other CV risk markers such as aortic pulse wave velocity (aPWV), validated predictive biomarkers of CV disease (NTproBNP, Troponin(I) hs), a promising CV biomarker (ST2 soluble) and coronary calcium score (CAC),
3. to study the association between asthma control and severity and various markers of CV risk.

To meet the study's objectives, volunteers from the EGEA study, recruited between 1991-95 in 5 centers (Paris, Grenoble, Lyon, Montpellier, Marseille) and who have not dropped out, will be contacted to take part in a new follow-up (EGEA4).

The new follow-up will consist of a clinical visit to :

* administer a standardized face-to-face (or postal) questionnaire similar to that used in previous EGEA surveys to assess respiratory and allergic symptoms and diseases, the presence of chronic comorbidities, including CV events (e.g. stroke, arteriosclerosis, heart attack), quality of life, asthma control, lifestyle, diet (using a validated food frequency questionnaire to assess average dietary intake over the past 12 months), social and environmental factors (e.g. smoking and indoor environment) ;
* perform a clinical examination including :

  * anthropometric measurements (height, weight, waist circumference and hip circumference) and impedance measurement
  * blood pressure measurements;
  * spirometry to measure pulmonary function;
  * a one-minute chair-lift test to assess functional capacity;
  * non-invasive measurement of an independent predictor of CV events, the aortic pulse wave velocity [aPWV], estimated by the speed of the pulse wave between the ankle and wrist;
* take a hair sample;
* take a blood sample; The visit will last 2h30 and will be carried out by clinical research staff trained in study procedures.

A second visit will be offered to volunteers at the Grenoble and Paris centers to take a non-invasive measurement assessed by CT scan (without injection), the Coronary Calcium Score (CAC), which is a predictor of the risk of cardiovascular events. If time permits, CAC can be measured during the first visit.

In addition, following the first visit, EGEA :

* equip the volunteer with an accelerometer (Actigraph). This accelerometer will be worn on the waist (or wrist) for one week;
* equip the volunteer with a passive pollution sensor (NO2). The volunteer will wear the sensor for one week. The sensor can be easily attached to a backpack/handbag.
* install the COBANET application on the volunteer's phone and explain how to use it. The purpose of this application is to collect information on the cleaning products used by the volunteer (product name and barcode), the frequency of use and the way in which these products are used (with or without protection, etc.);
* provide the volunteer with a kit containing the materials needed to collect stool samples
* create a "Nutrinet" account on the Nutrinet cohort platform, where the participant will log on in the days following the visit to complete three 24-hour dietary records.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in at least one of the previous EGEA surveys;
* to be affiliated to a social security scheme or to be a beneficiary of such a scheme.

Exclusion Criteria:

* Person deprived of liberty by judicial or administrative decision;
* Person subject to a legal protection measure (safeguard of justice, curatorship or guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Framingham score variability between asthmatics and non-asthmatics | during clinical examination
  The primary endpoint will be the variability of the Framingham score between asthmatics and non-asthmatics to assess the association between asthma and cardiovascular (CV) risk.

SECONDARY OUTCOMES:
Aortic pulse wave velocity | during clinical examination
  comparison of aortic pulse wave velocity between asthmatics and non-asthmatics
validated predictive biomarkers of CV disease (NTproBNP, Troponin(I) hs), | during clinical examination
  comparison of validated predictive biomarkers of CV disease (NTproBNP, Troponin(I) hs), between asthmatics and non-asthmatics
Soluble ST2 | during clinical examination
  comparison of a promising CV biomarker: soluble ST2 between asthmatics and non-asthmatics
coronary calcium score | during clinical examination
  comparaison du score calcique coronaire entre les asthmatiques et non asthmatiques

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Siroux, PHD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Hopital de la Croix Rousse, Lyon
  - APHM, Marseille
  - Hôpital Arnaud De Villeneuve, Montpellier
  - APHP - Hôpital Bichat Claude Bernard, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://cohorte-egea.fr/